CLINICAL TRIAL: NCT03955835
Title: Acandis Credo Intracranial Stent for Unsuccessful Recanalization After Thrombectomy (ACUTE)
Acronym: ACUTE
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: CREDO stent is now CE-marked for rescue stenting (new indication).
Sponsor: Acandis GmbH (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ACUTE
Record Dates: First submitted 2019-05-16; First posted 2019-05-20 (Actual); Last update posted 2021-10-21 (Actual); Status verified 2021-10

CONDITIONS: Acute Ischemic Stroke; Intracranial Stenosis
MeSH Terms: conditions — Ischemic Stroke | interventions — Therapeutics

STUDY DESIGN:
Intervention Model Description: Prospective, interventional treatment, single-arm, open-label, multi-centre trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- ACUTE (Other): Patients with acute ischemic stroke and proven large vessel occlusion (e.g. intracranial internal carotid artery or middle cerebral artery) with unsuccessful recanalization after endovascular treatment with mechanical thrombectomy and suspected underlying stenosis of the occluded intracranial artery amenable to stenting based on judgment by the treating neurointerventionalist.
  Interventions: Device: Treatment with Credo® stent together with the NeuroSpeed® PTA balloon catheter.

INTERVENTIONS:
Device: Treatment with Credo® stent together with the NeuroSpeed® PTA balloon catheter. — Self-expandable Credo® stent together with NeuroSpeed® PTA balloon catheter. Credo® and NeuroSpeed® are already CE approved products, for which within ACUTE an additional new indication shall be examined.

SUMMARY:
Study objective is to evaluate the efficacy and safety of acute permanent stenting of symptomatic intracranial stenosis following unsuccessful recanalization by thrombectomy in acute ischemic stroke with large vessel occlusion using the self-expandable Credo® stent together with the NeuroSpeed® PTA balloon catheter.

DETAILED DESCRIPTION:
Prospective, interventional treatment, single-arm, open-label, multi-center trial.

ELIGIBILITY:
Inclusion Criteria:

* Acute ischemic stroke from large vessel occlusion (LVO)
* Failed recanalization after treatment with thrombectomy, i.e. persistent occlusion of intracranial internal carotid artery (ICA), proximal segment (M1, M2) of the middle cerebral artery (MCA) (TICI 0-1)
* Small to moderate infarct core prior to initiation of thrombectomy (CT ASPECTS 6-10, DWI lesion < 70 ml)
* Suspected underlying stenosis of the occluded artery amenable to stenting by judgement of the treating neurointerventionalist
* Age 18- 80 years
* Informed consent (see below)
* Decision to perform angioplasty and stenting < 12 hours of symptom onset
* Previous passage of occlusion with microcatheter obtained

Exclusion Criteria:

* Large infarct core prior to initiation of thrombectomy (CT ASPECTS 0-5, DWI lesion > 70 ml)
* Vessel occlusion or stenosis of different known or suspected cause than atherosclerosis (e.g. vasculitis)
* Pre-stroke disability (MRS > 2)
* Any sign of intracranial haemorrhage on brain imaging prior to thrombectomy
* Any sign of intracranial vessel perforation during thrombectomy
* Contraindication against treatment with double anti-platelet treatment
* Current effective use of oral anticoagulants (e.g. INR > 1.7 for Vitamin K antagonists)
* More than 3 attempts for recanalization of target lesion prior to the use of the study device.
* Stenosis longer than the working length of the NeuroSpeed PTA balloon catheter.
* Diameter of the healthy vessel proximal and distal to the stenosis prevents save treatment with the NeuroSpeed PTA balloon catheter or is outside the indicated range of the Credo stent.
* Diameter of the target area is outside the indicated range of the Credo stent after predilation.
* Contraindication against anti-platelet or anticoagulation therapy
* Heavily calcified lesions that may prevent access or safe stent placement.
* Pregnant and breastfeeding women

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2019-08-09 (Actual); Primary Completion 2021-09-22 (Actual); Study Completion 2021-09-22 (Actual)

PRIMARY OUTCOMES:
Co-Primary Technical Efficacy Endpoint | Assessed after interventional procedure
  Technical success defined as successful recanalization of the occluded vessel (TICI 2b-3) at the end of the procedure (successful PTA + permanent stenting).
Co-Primary Clinical Efficacy Endpoint | 90 +/- 10 days after stroke
  Good clinical outcome 90 (±10) days after stroke defined as a score of 0-2 on the modified Ranking Score (MRS 0-2).
Primary Safety Endpoints | Within 18-36 hours after treatment
  * Symptomatic intracranial hemorrhage (SICH) as defined in SITS-MOST (within 18-36 hours of treatment)
  * Device-related procedural complications: Dissection, perforation or rupture of the target vessel, embolism, stent thrombosis or occlusion, stent migration.

SECONDARY OUTCOMES:
Secondary Efficacy Endpoints | 90 +/- 10 days after stroke
  * Categorical shift in MRS 90 (±10) days after stroke
  * Functional health status and quality of life 90 (±10) days after stroke (EQ-5D)
  * Infarct growth by 18-36 hours after stroke as compared to predicted infarct growth
  * Frequency of residual stenosis > 50 %
Secondary Safety Endpoints | 90 +/- 10 days after stroke
  * Ischemic stroke in downstream territory of the occluded vessel within 90 (±10) days after stroke
  * Parenchymal hemorrhage type 2 (PH-2) after 18-36 hours
  * Embolization in new territories
  * Mortality 90 (±10) days after stroke
  * Death or dependency 90 (±10) days after stroke (MRS 4-6)

CONTACTS AND LOCATIONS:
Locations (8):
- Germany (8):
  - Universitätsklinikum Hamburg-Eppendorf, Hamburg
  - Asklepios Klinik Altona, Abteilung für Radiologie und Neuroradiologie, Hamburg
  - Universitätsklinikum Heidelberg, Heidelberg
  - Klinik für Diagnostische und Interventionelle Neuroradiologie, Universitätsklinikum des Saarlandes, Homburg
  - Kliniken Maria Hilf GmbH Akademisches Lehrkrankenhaus der Uniklinik RWTH Aachen,Klinik für Diagnostische und Interventionelle Radiologie und Neuroradiologie, Mönchengladbach
  - Institut für Radiologie und Neuroradiologie, Evangelisches Krankenhaus Oldenburg, Oldenburg
  - Klinikum Osnabrück GmbH, Röntgen- und Strahlenklinik, Osnabrück
  - Abteilung für interventionelle Neuroradiologie, radprax an der St. Lukas Klinik, Solingen

IPD SHARING:
Plan to Share IPD: No